CLINICAL TRIAL: NCT07352787
Title: High-Intensity Laser Therapy for Trapezius Myofascial Pain Syndrome: Effects on Pain, ROM, Function, and Depression A Four-Phase Development, Validation, and Evaluation Study
Brief Title: High-Intensity Laser Therapy for Trapezius Myofascial Pain (HILT-TRAP Study)
Acronym: HILT-TRAP Stud
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neveen Abd El Maksoad Kohaf (Other)
Collaborators: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor-Investigator, Neveen Abd El Maksoad Kohaf, Clinical Pharmacy Department, Faculty of Pharmacy (Girls), Al-Azhar University, Cairo, Egypt., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HILT-TMPS-2026-4P-DEVVAL
Record Dates: First submitted 2026-01-04; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Myofascial Pain Syndrome (MPS)
Keywords: High-Intensity Laser Therapy; Trapezius Myofascial Pain Syndrome; Randomized Controlled Trial; Neck Pain; Physiotherapy
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Laser Therapy (HILT) (Experimental): Participants in this arm will receive active High-Intensity Laser Therapy applied to the trapezius muscle region for the treatment of trapezius myofascial pain syndrome.
  Interventions: Device: High-Intensity Laser Therapy
- Sham Laser Therapy (Placebo Comparator): Participants in this arm will receive sham laser therapy applied to the trapezius muscle region. The sham procedure will mimic the appearance and application of active laser therapy without delivering therapeutic laser energy.
  Interventions: Device: Sham Laser Therapy

INTERVENTIONS:
Device: High-Intensity Laser Therapy — High-Intensity Laser Therapy will be administered using a class IV therapeutic laser device applied over identified trapezius myofascial trigger points and surrounding muscle tissue. Treatment parameters (wavelength, power output, energy density, and duration) will follow standardized clinical protocols and safety guidelines. Sessions will be delivered by a licensed physical therapist, with participants receiving multiple treatment sessions over the intervention period. The therapy aims to promote analgesia, improve microcirculation, reduce muscle tension, and facilitate tissue healing.
  Arms: High-Intensity Laser Therapy (HILT)
Device: Sham Laser Therapy — Sham laser therapy will be administered using an identical laser device and treatment procedure; however, no therapeutic laser energy will be emitted. The duration, frequency, and therapist interaction will be identical to the active treatment.
  Arms: Sham Laser Therapy

SUMMARY:
This study aims to evaluate the effectiveness of optimized High-Intensity Laser Therapy (HILT) compared with sham treatment in patients with trapezius myofascial pain syndrome. Outcomes include pain intensity, cervical range of motion, functional disability, and depressive symptoms measured at baseline, post-intervention, and 16-week follow-up.

DETAILED DESCRIPTION:
Myofascial pain syndrome of the trapezius muscle is a common cause of chronic neck and shoulder pain associated with functional limitation and psychological distress. Although High-Intensity Laser Therapy is increasingly used in clinical practice, high-quality evidence regarding its long-term effects and optimal treatment parameters is limited.

This double-blind, randomized, placebo-controlled trial will enroll 104 adults with clinically diagnosed trapezius myofascial pain syndrome. Participants will be randomly assigned to receive either optimized High-Intensity Laser Therapy or sham laser treatment. Outcomes will be assessed at baseline, immediately after the intervention, and at 16-week follow-up. This study aims to provide evidence for a standardized, patient-centered HILT protocol suitable for routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Clinically diagnosed trapezius myofascial pain syndrome
* Duration of symptoms ≥ 4 weeks
* Pain intensity ≥ 4 on NPRS
* Able to provide informed consent

Exclusion Criteria:

* Red-flag medical conditions (e.g., malignancy, spinal cord compression)
* Neurological disorders affecting the neck or shoulder
* Cognitive impairment or inability to communicate
* Previous laser therapy to the neck/shoulder region within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-03-10 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 16-week follow-up
  Pain intensity will be evaluated using the Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable.

SECONDARY OUTCOMES:
Functional Disability | 16-week follow-up
  Neck Disability Index (NDI)
Cervical Range of Motion | 16-week follow-up
  Measured using CROM device
Depression | 16-week follow-up
  Beck Depression Inventory-II (BDI-II)

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Hussein Teaching Hospital, Nasiriyah, Nasiriyah, Iraq

IPD SHARING:
Plan to Share IPD: No